CLINICAL TRIAL: NCT00224497
Title: A Phase IIa/b Double-blind, Randomised, Placebo-controlled, Linear Trend Design Dose-ranging Study to Investigate the Effects of 24 Weeks of Monotherapy With SB-742457 on Cognition in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Dose Ranging Study To Investigate The Efficacy And Safety Of SB-742457 In Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ3100603
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; cognition global functioning; symptomatic; B-742457
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

INTERVENTIONS:
Drug: SB-742457

SUMMARY:
The purpose of this study is to find out if SB-742457 is a safe treatment and what effects it has on the symptoms of mild to moderate Alzheimer's disease. SB-742457 is a new treatment which is thought to increase the levels of certain chemicals in the brain that are often decreased in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of probable mild-to-moderate Alzheimer's disease as determined by the NINCDS-ADRDA and DSM-IV criteria with an MMSE score of 12-24.
* Subjects and their caregivers must provide informed consent prior to study entry.
* Adequate blood pressure and laboratory values.

Exclusion criteria:

* Females of child-bearing potential.
* Have other causes of dementia such as vascular damage, depression, bipolar affective disorder, schizophrenia, syphilis, vitamin B12 deficiency or thyroid deficiency.
* Subjects taking medication for Alzheimer's disease or centrally acting agents which might impact study outcomes.
* Subjects taking agents for which there is a theoretical risk of interaction with SB-742457.
* Subjects with known hypersensitivity to sunlight or seizures.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-09

PRIMARY OUTCOMES:
Change in cognition and function after 24 weeks.

SECONDARY OUTCOMES:
Change in behavioural symptoms, activities of daily living and caregiver burden after 24 weeks. Changes in all symptoms at 8 and 12 weeks. Safety and tolerability. PK and dose response profiling. Efficacy related to ApoE status.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (37):
- Austria (4):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Retz
  - GSK Investigational Site, Vienna
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Croatia (2):
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Czechia (4):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rychnov nad Kněžnou
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
- Poland (3):
  - GSK Investigational Site, Mosina
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Rimavská Sobota
- South Africa (3):
  - GSK Investigational Site, Oakdale
  - GSK Investigational Site, Rosebank
  - GSK Investigational Site, Somerset West
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sant Cugat Del Vallés/
  - GSK Investigational Site, Tarrasa, Barcelona